CLINICAL TRIAL: NCT03986931
Title: A Pharmacist Intervention for Monitoring and Treating Hypertension Using Bidirectional Texting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linnea Polgreen (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Linnea Polgreen, Associate Professor, Department of Pharmacy Practice and Science / Division of Health Services Research, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BP Texting and Pharmacist; R61HL144880 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Research interns conducting baseline and exit data collection will be blinded so that they do not influence responses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-Bidirectional Texting Group (Experimental): Patients enrolled in the Pharmacist-Bidirectional Texting Group will return 7 morning and 7 evening blood pressure measurements via text message. The report will be shared with a pharmacist who will monitor them for 12 months. The pharmacist will have access to their entire medical record and will provide support and education via text messaging, email, or phone calls, whichever is preferred by the patient. The pharmacist will develop a care plan and make recommendations to the physician through the electronic medical record to quickly adjust therapy to improve control. They will also recommend laboratory testing if indicated. They will have contact with the patient every 2-3 weeks while blood pressure is uncontrolled, and at least every 2 months when it is controlled. The pharmacist will track all recommendations made to physicians and whether or not they were implemented, modified, or rejected.
  Interventions: Other: Experimental: Pharmacist-Bidirectional Texting Group
- Control Group (Active Comparator): Patients randomized to the control group will also return 7 morning and 7 evening blood pressure measurements. The report will be shared with a pharmacist who will call the patient to discuss the measurements and possibly recommend follow up with a physician, but no other pharmacist intervention or monitoring will occur during the 12 months.
  Interventions: Other: Active Comparator: Control Group

INTERVENTIONS:
Other: Experimental: Pharmacist-Bidirectional Texting Group — The goal of this intervention is to determine if bidirectional texting and pharmacist monitoring will improve blood pressure control.
  Arms: Pharmacist-Bidirectional Texting Group
Other: Active Comparator: Control Group — This group will receive bidirectional texting, but no pharmacist monitoring.
  Arms: Control Group

SUMMARY:
Bidirectional texting is an effective way to collect home blood pressure (BP) measurements from subjects, but collecting BP measurements and sending them to physicians does not necessarily lead to decreased BP. Pharmacist interventions have been successful in decreasing subject BP. However, pharmacists are expensive, and in successful interventions, spent a substantial amount of time collecting home BP measurements. In this study, a proven pharmacist intervention will be added to a bidirectional texting program to determine if a combined pharmacist-bidirectional texting intervention is successful at decreasing subject BP and increasing subject BP treatment intensification in a cost-effective manner. This study will be a cluster-randomized, controlled trial of a new intervention.

DETAILED DESCRIPTION:
HTN is associated with the greatest attributable risk for mortality among all modifiable risk factors for cardiovascular disease.[1] In 2014, there were approximately 72 million adults (29%) with HTN in the US.[2] Several clinical trials have demonstrated that antihypertensive medications reduce cardiovascular events.[3] For example, even a 5 mm Hg difference in systolic BP (SBP) over 3-5 years can reduce the risk of cardiovascular complications and strokes by 25-30%.[4] Yet, approximately 20% of U.S. adults are unaware of their HTN,[5] and among patients diagnosed with HTN, 47% are uncontrolled.[2] Thus, there is a critical need to effectively treat patients with HTN.

Clinical inertia has been identified as the primary cause for delays in achieving BP control for over 20 years.[6-8] Providers often discount office BP readings that may be falsely elevated due to observer or measurement error and/or the clinical surroundings (e.g., white coat HTN).[9-11] Patients are often seen only once or twice a year which further delays BP control. Furthermore,[8, 12] BP goals are achieved in only 49% of the patients who take anti-hypertensive medications.[5] New approaches for acquiring more BP readings are also needed to better monitor and titrate treatment because a significant proportion of patients on therapy are not adequately controlled despite frequent physician visits.

Home BP measurements, (i.e., having patients take their BP at home), can facilitate the more timely diagnosis of HTN by reducing diagnostic uncertainty. In fact, home measurements are better prognostic indicators of stroke and cardiovascular mortality than clinic measurements,[13-15] are more closely correlated with end-organ damage from HTN than clinic measurements,[16, 17] are cost effective and well-tolerated by patients,[18] and generate BP readings that are at least as reproducible as clinic readings.[19] Home BP measurements, if available, may help physicians overcome barriers related to clinical inertia.[20] However, the data must be followed by action. The researchers have pioneered physician-pharmacist collaborative management (PPCM) that has been shown to decrease clinical inertia and improve BP control.[21, 22] Pharmacists have been embedded within the medical office to perform BP management. The pharmacists are able to assess patients' needs and provide recommendations to physicians regarding treatment changes, providing patients with timely therapy adjustments.[23] However, many medical office leaders are unable to hire clinical pharmacists due to limited resources. Therefore, a "virtual", remote clinical pharmacy service has been developed.[24] Pharmacists were able to obtain electronic medical record (EMR) access at all intervention offices for private physician offices throughout Iowa. While the physicians accepted 95% of the pharmacists' recommendations, the effect on improving BP was modest (manuscript under review). Adding the proposed texting platform with home BP monitoring should markedly improve the potency of our remote, telepharmacy intervention.

This trial exhibits clinical equipoise because, although it is known that texting is an efficient method for obtaining home BP measurements, and that pharmacist interventions to improve BP are cost-effective, it is not known if combining these two interventions will also be cost effective. There are four reasons why this study might not be successful. First, while meta-analyses have found significantly improved BP with pharmacist interventions some studies were not successful.[25] Second, more data does not necessarily mean better data: patients could report false values, BP could be abnormally low or high during the measurement period, or the data could be ignored. Third, even better data might not lead to better outcomes: data could be ignored by pharmacists, physicians or patients; pharmacists' recommendations could be ignored by physicians or patients. Fourth, even if the study is effective at improving subject outcomes, it might not be cost effective. Texting might not save as much time as hypothesized. Thus, further research is needed to address these gaps in knowledge.

There is a critical need for an easy-to-use, cost-effective, mobile health (m-health) approach to assist patients and healthcare providers with screening, diagnosis, and monitoring of HTN. Small medical offices and those located in poor or rural areas are unable to operationalize team-based care with pharmacists. The researchers have overcome this barrier with the use of a remote clinical pharmacy services. Coronary heart disease deaths could be reduced by 15-20% and stroke deaths by 20-30% if this intervention effectively improves BP and is implemented more widely in primary care offices.

The goal of this proposal is to evaluate whether a scalable, short messaging service (SMS) approach combined with a pharmacist-based intervention improves BP management cost effectively. To achieve this objective, the following specific aims are proposed:

1. Determine if mean BP 12 months after the intervention decreases more for the intervention group than the control group. The working hypothesis is that those in the pharmacist-intervention group will achieve larger BP decreases than those in the control group.
2. Determine if the intervention leads to more intensification of therapy than in the control group. The working hypothesis is that subjects in the pharmacist-intervention group will have more treatment changes than those in the control group.
3. Determine the cost effectiveness of the intervention. The working hypothesis is that the intervention will be cost effective when compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English or Spanish
* Have a clinic measured blood pressure of > or = 145 mmHg and/or > or = 95 mmHg at two previous clinic visits or one previous clinic visit and on the day of enrollment
* Must be a patient at Family Medicine, River Crossings, Scott Blvd, or Muscatine University of Iowa Clinics
* Live in a zip code that is scored as a 4-10 on the Rural-Urban Commuting Area codes

Exclusion Criteria:

* Currently pregnant or planning to become pregnant in the next year
* Upper arm circumference greater than 50 cm (20 in)
* Prisoner status
* Unable to provide own informed consent

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linnea A Polgreen, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Polgreen LA, Carter BL, Polgreen PM, Snyder PM, Sewell DK, Bayman EO, Francis SL, Simmering JE, Parker C, Finkelstein R. A pharmacist intervention for monitoring and treating hypertension using bidirectional texting: PharmText BP. Contemp Clin Trials. 2020 Nov;98:106169. doi: 10.1016/j.cct.2020.106169. Epub 2020 Oct 7. PMID 33038500

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant must have an average research blood pressure > 145 mmHg systolic or > 95 mmHg diastolic measured by a research team member on the day of enrollment to be eligible to continue participation.
  535 participants signed a consent form. 114 participants did not pass the additional blood pressure screening and were not randomized. 1 participant died prior to randomization. 420 participants were randomized.
Period: Overall Study
Arm/Group | Pharmacist-Bidirectional Texting Group | Control Group
Started | 209 | 211
Completed | 209 | 211
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist-Bidirectional Texting Group | Control Group | Total
Number analyzed (Participants) | 209 | 211 | 420
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (13.7) | 58.4 (13.6) | 58.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 113 | 209
  Male | 113 | 98 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 48 | 97
  Not Hispanic or Latino | 160 | 162 | 322
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 5 | 16
  White | 184 | 196 | 380
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 7 | 9 | 16
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Body mass index (BMI) missing for 4 participants in Intervention group and 8 participants in the Control group.
  kg/m^2 | 32.6 (7.4) | 33.7 (7.8) | 33.1 (7.7)
Level of Education [Count of Participants; unit: Participants]
  < High School | 32 | 46 | 78
  High School | 66 | 56 | 122
  Some College | 37 | 46 | 83
  Associate's Degree | 27 | 20 | 47
  Bachelor's Degree | 30 | 24 | 54
  Master's Degree | 10 | 10 | 20
  Doctoral Degree | 5 | 6 | 11
  Trade School | 2 | 3 | 5
Smoking History [Count of Participants; unit: Participants]
  Never Smoked | 117 | 120 | 237
  Current Smoker | 37 | 34 | 71
  Former Smoker | 55 | 57 | 112
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 156.0 (13.7) | 153.4 (14.0) | 154.3 (14.0)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 88.4 (12.3) | 90.1 (12.5) | 89.5 (11.9)
10-Year Atherosclerotic Cardiovascular Disease (ASCVD) Risk [Mean (Standard Deviation); unit: Percentage] — The ASCVD risk score is given as a percentage. This is your chance of having heart disease or stroke in the next 10 years. Individuals are preliminarily classified based on estimated risk: 10-year ASCVD risk <5% is low risk; 5%-7.5% is borderline risk; 7.5-20% is intermediate risk, and ≥20% is high risk. Population: Many variables are required to calculate an ASCVD Risk Score. If any variables are missing, the score cannot be calculated.
  Percentage
    number analyzed (Participants) | 89 | 109 | 198
    (all) | 17.3 (14.2) | 15.0 (14.7) | 16.0 (14.5)
Medical History [Number; unit: participants]
  Angina | 22 | 8 | 30
  Chronic Kidney Disease | 13 | 11 | 24
  Coronary Artery Disease | 18 | 12 | 30
  Diabetes Mellitus | 57 | 65 | 122
  Heart Failure | 10 | 6 | 16
  Hyperlipidemia | 60 | 53 | 113
  Heart Attack | 10 | 4 | 14
  Stroke | 11 | 5 | 16
  Transient Ischemic Attack (TIA) | 1 | 2 | 3
Hypertension Medications [Mean (Standard Deviation); unit: medications] | 1.7 (1.2) | 1.5 (1.3) | 1.6 (1.2)
Rural-Urban Commuting Area Codes [Count of Participants; unit: Participants] — The USDA Economic Research Service developed the rural-urban commuting area (RUCA) codes to classify U.S. regions as rural/urban using measures of population density, urbanization, and daily commuting. Lower RUCA scores indicate that a participant lives in a more urban area, whereas higher RUCA scores indicate that the participant lives in a more rural area. Participants must have a RUCA code >= 4 to be eligible for the study since our focus was on monitoring blood pressure in rural participants.
  Participants
    RUCA 4 | 35 | 44 | 79
    RUCA 5 | 21 | 15 | 36
    RUCA 6 | 1 | 0 | 1
    RUCA 7 | 80 | 73 | 153
    RUCA 8 | 5 | 2 | 7
    RUCA 9 | 3 | 5 | 8
    RUCA 10 | 64 | 72 | 136

OUTCOME MEASURES:

1. Primary Outcome: Difference in Change in Systolic Blood Pressure- 12 Months
Description: The difference between the groups in the change from baseline to 12 months in systolic blood pressure in mm Hg.
Time Frame: 12 months
Population: Blood pressure was measured by the research team at baseline, 6 months, and 12 months. All participants had a baseline measurement. Some were missing 6- or 12-month measurements. All collected measurements were included in the model estimation.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: BP Measurements
Arm/Group | Pharmacist-Bidirectional Texting Group | Control Group
Number analyzed (Participants) | 209 | 211
Number analyzed (BP Measurements) | 494 | 511
mmHg | -23.8 (19.4) | -19.6 (19.4)

2. Secondary Outcome: Difference in Change in Diastolic Blood Pressure- 12 Months
Description: The difference between the groups in the change from baseline to 12 months in diastolic blood pressure in mmHg.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: BP Measurements
Arm/Group | Pharmacist-Bidirectional Texting Group | Control Group
Number analyzed (Participants) | 209 | 211
Number analyzed (BP Measurements) | 494 | 511
mmHg | -9.1 (13.4) | -9.6 (11.4)

3. Secondary Outcome: Number of Medication Changes From 6 to 12 Months
Description: Total number of medication changes (i.e., dose, discontinuation, initiation, etc.) from 6 months to 12 months as documented in the medical record.
Time Frame: 12 months
Population: All participants had a BP medication chart review at baseline, 6 months, and 12 months unless they withdrew from the study prior to a chart review period.
Measure: Mean (Standard Deviation); unit: Medication Changes
Units Other Than Participants: Medication Chart Reviews
Arm/Group | Pharmacist-Bidirectional Texting Group | Control Group
Number analyzed (Participants) | 209 | 211
Number analyzed (Medication Chart Reviews) | 392 | 405
Medication Changes | 0.59 (0.98) | 0.44 (0.84)

4. Secondary Outcome: Dollars Spent Per Patient for 12 Month Bidirectional Texting/Pharmacist Intervention
Description: Total cost of medications, time spent by research staff, and clinics visits per patient from baseline.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Pharmacist-Bidirectional Texting Group | Control Group
Number analyzed (Participants) | 209 | 211
Dollars | 980.17 (1127.91) | 838.95 (713.45)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Pharmacist-Bidirectional Texting Group | Control Group
All-Cause Mortality (participants affected / at risk) | 7/209 | 4/211
Serious Adverse Events (participants affected / at risk) | 0/209 | 0/211
Other Adverse Events (participants affected / at risk) | 0/209 | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT03986931/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03986931/ICF_001.pdf